CLINICAL TRIAL: NCT06137313
Title: Determination of HEV Seroprevalence Among Blood Donors in Occitania
Brief Title: Exposure to Hepatitis E Virus in Occitania, France
Acronym: EVE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0505
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hepatitis E
MeSH Terms: conditions — Hepatitis E | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — completion of a questionnaire

SUMMARY:
The objective of the proposed work is to determine the seroprevalence of HEV in 2023 in a population of blood donors living in Occitania.

Compare the current frequency of anti-HEV IgG and IgM markers with that of 2011. The serological techniques used and the questionnaires will be similar

DETAILED DESCRIPTION:
Hepatitis E virus (HEV) includes 4 major genotypes. It is now well established that HEV is endemic in most industrialized countries where it is transmitted zoonotically (genotypes 3 and 4) from a large animal reservoir, mainly pigs, unlike in resource-limited countries where it is is transmitted by water (genotypes 1 and 2 strictly human). The optimization of the use of virological tests and the improvement of epidemiological knowledge have led to the identification of a growing number of hepatitis E transmitted enterically but also through transfusion. While many infections are asymptomatic and self-limiting, immunocompromised people can develop chronic hepatitis which can progress to cirrhosis. Furthermore, people with pre-existing chronic hepatitis regardless of the etiology present, in the event of HEV infection, a risk of hepatic decompensation associated with high mortality. The diagnosis of HEV infection is based on both serological tests (anti-HEV IgM and anti-HEV IgG) and molecular tests (HEV RNA).

Although HEV transmission is mainly enteric, transmission by labile blood products (plasma, platelets, or red blood cells) has been documented in France and abroad. Given the endemic nature of HEV infection on a global scale and the very high frequency of asymptomatic infections, reducing the risk of HEV transmission by transfusion cannot be achieved by selecting donors from clinical or epidemiological criteria. Furthermore, pathogen mitigation processes are ineffective on HEV. As a result, biological screening for HEV has been implemented in different countries in Europe and Asia. In France, systematic screening of the HEV genome was introduced on March 20, 2023. All positive samples are sent to the HEV-hepatitis A virus (HAV) National Reference Center (Toulouse University Hospital Virology Laboratory) for quantification of the viral load, determination of the genotype and detection of anti-HEV antibodies (IgG and IgM). Donors screened positive for HEV-RNA are informed of the infection by a specific letter and invited to consult a General Practitioner. Hygiene measures are also recommended to prevent contamination of those around you due to viral excretion in the stools. They are deferred from donating for a period of 4 months corresponding to a maximum duration of viremia. An epidemiological questionnaire is completed by the donor and returned by mail to the French Blood Establishment.

Previous studies conducted more than 10 years ago among blood donors in Occitanie and at the national level showed that the Occitanie region was a region with high HEV seroprevalence (39%) but with differences ranging from 20% to more than 70% depending on the departments. Based on multivariate analyses, dietary habits such as consumption of pork or game do not explain the entire epidemiology of HEV in this region and other modes of transmission, notably by water, probably exist.

ELIGIBILITY:
Inclusion Criteria:

* blood donors

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult blood donors
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of blood donors harbouring IgG anti-HEV | at inclusion
  analysis of IgG anti-HEV in serum

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Izopet, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No